CLINICAL TRIAL: NCT03144778
Title: Checkpoint Inhibitors Assessment in Oropharynx Carcinoma (CIAO)
Brief Title: Durvalumab With or Without Tremelimumab in Treating Participants With Stage II-IVA Oropharyngeal Squamous Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0805; NCI-2018-01199 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0805 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Stage II Oropharyngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (durvalumab) (Experimental): Participants receive durvalumab IV over 1 hour on days 1 and 29 in the absence of disease progression or unaccepted toxicity. Between days 52 and 72, participants undergo standard of care surgery.
  Interventions: Biological: Durvalumab
- Cohort II (durvalumab, tremelimumab) (Experimental): Participants receive durvalumab IV over 1 hour and tremelimumab IV over 1 hour on days 1 and 29 in the absence of disease progression or unaccepted toxicity. Between days 52 and 72, participants undergo standard of care surgery.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
  Arms: Cohort II (durvalumab, tremelimumab)

SUMMARY:
This phase I trial studies how well durvalumab with or without tremelimumab works in treating participants with stage II-IVA oropharyngeal squamous cell cancer. Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the differences between CD8+ tumor infiltrating lymphocytes evaluated by immunohistochemistry staining in the post-treatment surgical specimens as compared to baseline in patients treated with durvalumab single agent compared with patients receiving durvalumab plus tremelimumab.

SECONDARY OBJECTIVES:

I. Safety and toxicity of durvalumab single agent or combined with tremelimumab administered every 4 weeks for 2 doses in the preoperative setting according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

II. Objective Response rate at 8 weeks, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

III. Percentage of patients undergoing the initially proposed surgery at 4 weeks.

IV. Percentage of patients undergoing the initially proposed surgery at 8 weeks.

V. Percentage of viable tumor cells in the surgical specimen. VI. Patient-reported outcomes (PRO) during treatment with checkpoint inhibitors.

EXPLORATORY OBJECTIVES:

I. To assess pre- and post- treatment tumor, blood and oral rinse based immune biomarkers.

II. Correlate tissue and blood-based biomarkers with human papillomavirus (HPV) status, outcomes and toxicity.

OUTLINE: Participants are randomized into 1 of 2 cohorts.

COHORT I: Participants receive durvalumab intravenously (IV) over 1 hour on days 1 and 29 in the absence of disease progression or unaccepted toxicity. Between days 52 and 72, participants undergo standard of care surgery.

COHORT II: Participants receive durvalumab IV over 1 hour and tremelimumab IV over 1 hour on days 1 and 29 in the absence of disease progression or unaccepted toxicity. Between days 52 and 72, participants undergo standard of care surgery.

After completion of study treatment, participants are followed up at 28 and 42 days, 4 and 6 months, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study according to the investigational review board (IRB)
* Suspected or histologically/cytologically confirmed oropharyngeal squamous cell carcinoma (OPSCC), stage II, III, or IVA (according to the American Joint Committee on Cancer [AJCC] 7th edition), or patients with loco-regional recurrence from an OPSCC primary, if time of recurrence is at least 6 months after completion of initial curative intent treatment (surgery or radiotherapy +/- chemotherapy or cetuximab). Patients with a suspected lesion may be enrolled and a baseline biopsy will be obtained as part of the study. If squamous cell histology is not confirmed, patients will be discontinued from the study
* Patients must have surgically resectable disease in the opinion of the treating physician. For patients with a primary OPSCC, patients must be eligible for TORS (transoral robotic surgery)
* Available tissue from prior biopsy (minimum of 10 unstained slides), or willing to undergo core biopsy to obtain tumor material. Biopsy will be mandatory for patients with recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (> 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula
* Patients with reproductive potential (e.g., females menopausal for less than 1 year and not surgically sterilized) must practice two highly effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of durvalumab monotherapy or for at least 180 days after completion of durvalumab/tremelimumab combination therapy. Female patients of childbearing potential must provide a negative pregnancy test (urine) prior to treatment initiation
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Histology other than squamous cell carcinoma
* Primary site other than oropharynx
* Prior systemic therapy (chemotherapy, biologic, or immunotherapy) for the same OPSCC. Prior chemotherapy, biologic therapy, and radiotherapy is allowed in patients with loco-regional recurrent disease, if administered at least 6 months prior to study enrolment
* Previous treatment with Anti-CTLA-4 including tremelimumab or PD1/PD-L1 inhibitor, including durvalumab
* History of another primary malignancy except for: (i) OPSCC with loco-regional recurrence after 6 months of curative-intent treatment and amenable to salvage surgery; (ii) malignancy treated with curative intent and with no evidence of active disease >= 2 years before the first dose of study drug and of low potential risk for recurrence; (iii) non-melanoma, skin cancer or lentigo maligna; in situ cervical, breast, prostate or bladder carcinoma
* Any concurrent anticancer therapy
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from a baseline electrocardiogram using Fridericia's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, and single dose of dexamethasone of up to 20 mg (or equivalent corticosteroid) administered prior to diagnostic or baseline study biopsy of the oropharynx, as per institution standard of care
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or pneumonitis
* History of primary immunodeficiency
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, seizures, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of active tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing two highly effective methods of birth control
* Any medical or psychosocial condition that will interfere with evaluation of study treatment or interpretation of patient safety or study results
* Known allergy or hypersensitivity to investigational product (IP) or any excipient
* Any unresolved grade 2 or higher toxicity from previous anti-cancer therapy
* Primary tumor not amenable to TORS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change of CD8+ tumor infiltrating lymphocytes | Before and after treatment, assessed up to 5 years
  Change will be defined as the ratio of the CD8+ lymphocytes density in the post-treatment surgical specimens over the CD8+ density in the baseline biopsy before treatment.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | Up to 5 years
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.
Overall response rate | At 8 weeks
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1.
Mean MD Anderson Symptom Inventory Head and Neck Cancer (MDASI-HN) | At 29 Days
  The Mean MD Anderson Symptom Inventory Head and Neck Cancer (MDASI-HN) is a 28-item patient-reported outcomes questionnaire developed to measure severity or burden of systemic and head and neck squamous cell carcinoma (HNSCC)-specific symptoms and their interference with patients' daily functioning. Each symptoms is rated from 0 (not present) to 10 (as bad as you can imagine).
Percentage of viable tumor cells in the surgical specimen | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ferrarotto R, Bell D, Rubin ML, Hutcheson KA, Johnson JM, Goepfert RP, Phan J, Elamin YY, Torman DK, Warneke CL, Hessel AC, Garden AS, Myers JN, Johnson FM, Lee JJ, Sikora AG, Gillison ML, Glisson BS, Gross ND. Impact of Neoadjuvant Durvalumab with or without Tremelimumab on CD8+ Tumor Lymphocyte Density, Safety, and Efficacy in Patients with Oropharynx Cancer: CIAO Trial Results. Clin Cancer Res. 2020 Jul 1;26(13):3211-3219. doi: 10.1158/1078-0432.CCR-19-3977. Epub 2020 Apr 8. PMID 32269052
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org